CLINICAL TRIAL: NCT02809885
Title: Hepatitis E Virus Infection in Pediatric Transplantation, a Prevalence Study
Acronym: HEV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2013-810
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Transplantation
Keywords: Hepatitis E; Pediatric; Transplantation; Prevalence
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transplanted patients (Experimental): All patients included are in the same arm.
  Interventions: Biological: Hepatitis E serology

INTERVENTIONS:
Biological: Hepatitis E serology

SUMMARY:
Hepatitis E virus (HEV) is an emerging disease. The genotype 1 and 2 are predominant in Asia and Africa, and are responsible for recurrent epidemics. Genotype 3 is the main genotype found in Europe and North America and is responsible for sporadic infections except for travel associated diseases.

HEV had a principally asymptomatic form. However, it was recently demonstrated that it could lead to a chronic form, especially in immunosuppressed patients. Moreover, in liver transplanted patients the infection could mimic a rejection and lead to the loss of the transplant. In other immunosuppressed patients, chronic hepatitis lead to cirrhosis and its well-known complications (ascitis, digestive hemorrhage, liver failure...). There is a lack of information about the prevalence of this disease.

In Canada the incidence of HEV infection was high (15-86% for liver transplanted children with liver tests disturbed). In Germany the prevalence was lower: 3,2% in liver & kidney transplanted children whereas 7,4% in control. It was shown in a retrospective study that in liver (and liver+kidney) transplanted children the prevalence in Lyon was around 8,3%.

This study will determined in a prospective approach the HEV prevalence in kidney, lung, heart and bone marrow transplanted children in Lyon.

ELIGIBILITY:
Inclusion Criteria:

* <18 years old
* transplantation (heart, kidney, lung or bone marrow)
* protocol acceptance by family
* social security available

Exclusion Criteria:

* protocol rejection by family

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 226 (Estimated)
Dates: Start 2013-12-19 (Actual); Primary Completion 2017-12-19 (Estimated); Study Completion 2017-12-19 (Estimated)

PRIMARY OUTCOMES:
Hepatitis E virus prevalence in pediatric transplanted patients | Day 1
Hepatitis E virus prevalence in pediatric transplanted patients | 6 months
  Hepatitis E virus (HEV) serology : IgG & IgM, and PCR HEV. If serology is positive a second serology will be performed 6 months after in order to detect chronic infection.

SECONDARY OUTCOMES:
Correlation between HEV prevalence and the different types of transplantation | Day 1
Correlation between HEV prevalence and the different types of transplantation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No